CLINICAL TRIAL: NCT05955612
Title: Use of Procalcitonin Point-of-care Test to Guide De-escalation of Empiric Antibiotic Therapy in Adult Patients With Sepsis in a Tertiary Hospital in Bangladesh (PROCALBAN): a Phase 3 Randomised, Controlled, Open-label Trial
Brief Title: Use of Procalcitonin, a Blood Test to Guide Antibiotic Therapy for Sepsis in Adults
Acronym: PROCALBAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BAC23002
Record Dates: First submitted 2023-06-22; First posted 2023-07-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Procalcitonin

STUDY DESIGN:
Masking Description: Procalcitonin measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily measurement of serum procalcitonin concentrations (Experimental)
  Interventions: Procedure: Procalcitonin measurement
- Standard of practice (routine clinical care) (No Intervention)

INTERVENTIONS:
Procedure: Procalcitonin measurement — Daily measurement of serum procalcitonin concentrations to guide de-escalation of antibiotics
  Arms: Daily measurement of serum procalcitonin concentrations

SUMMARY:
Trial design:

Randomised controlled, two-arm, parallel, clinical trial to assess the efficacy and safety of sequential daily procalcitonin assessments to guide de-escalation of empirical antibiotic therapy in adult patients with sepsis.

Trial settings Trial site is Chattogram Medical College Hospital (CMCH), Bangladesh. CMCH is tertiary care hospital with undergraduate and postgraduate teaching facilities. This tertiary hospital receives referrals from urban and rural areas of southern Bangladesh and has basic facilities for intensive care and haemodialysis.

Trial Participants:

Male or female hospitalised patients, 16-65 years of age, with confirmed or suspected sepsis Patients (Total 532) will be 1:1 randomised to either:

* Intervention arm: daily measurement of serum procalcitonin concentrations to guide de-escalation of antibiotics (Intervention arm: 266), or
* Control arm: standard of practice to guide de-escalation of antibiotics without procalcitonin assessments (Control arm: 266).

Patients will be followed-up until ICU discharge and/or hospital discharge with an additional follow-up at 28 days after discharge.

Funder: Wellcome Trust of Great Britain

Grant reference number from Wellcome Trust: 220211/A/20/Z

ELIGIBILITY:
Inclusion Criteria:

* Participant, legally authorised person/ legal guardian willing and able to give informed consent for participation in the trial.
* Male or Female, aged 16 to 65 years
* Suspected or proven bacterial infection
* A positive sepsis screening National Early Warning Score (NEWS) equal or greater than 5 (Table 1 or at least one criterion with a score of 3.
* Intention to start parenteral antibiotic therapy
* Within 24 hours of hospital admission

Exclusion Criteria:

* Patients with suspected/documented tuberculosis, parasitic infection (including malaria or visceral leishmaniasis), or viral infections (i.e., COVID-19, dengue, HIV)
* Pregnancy
* Intended for a short stay in ICU or general ward (such as post-operative)
* Patients requiring a predefined long course of antibiotic therapy (such as endocarditis, osteomyelitis, lung abscess, liver abscess, septic arthritis)
* Immunocompromised patients, including as severe neutropenia (< 500 cells/ml), transplant recipients, on prolonged corticosteroid treatment, chemotherapy or disease modifying immunomodulatory medications
* More than 48 hours of parenteral antibiotic use
* Surgical patients, including patients with a surgical septic source or patients requiring source control, i.e. abscess drainage
* Moribund patients or patients receiving end of life care
* Previous enrolment in PROCALBAN
* Conditions accompanied with a systemic inflammatory state, including pancreatitis, cardiogenic shock, severe trauma

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Length of antibiotic treatment | Through study completion, an average of 1 month
  number of days of antibiotic treatment during the study period.

SECONDARY OUTCOMES:
Consumption of antibiotics expressed as the Defined Daily Dosage (DDD) | Through study completion, an average of 1 month
  Defined daily dose (DDD) is the assumed average maintenance dose per day for a drug used in its main indication in adults.
Days of therapy with antibiotics (DOT) | Through study completion, an average of 1 month
  Definition of DOT: One DOT represents the administration of a single antibiotic on a given day regardless of the number of doses administered or dosage strength. If a patient receives more than one antibiotic it will be added on with DOT of the first antibiotic.
Number of days of parenteral antibiotic during hospitalisation period | Through study completion, an average of 1 month
  Number of days of parenteral antibiotic from the day of enrolment to the day of stopping of parenteral antibiotic during hospitalisation period
Number of days of antibiotic treatment during the hospitalisation period. | Through study completion, an average of 1 month
Overall mortality, mortality associated with recurrent infection and non-lethal recurrent infections. | Through study completion, an average of 1 month
  Recurrent infections are classified as follows: culture-positive relapse (unsuccessful eradication of the original infecting strain), culture-negative relapse (reappearance of symptoms after antibiotics cessation with negative cultures), reinfection (infection by a different strain of the same species), and syndromic recurrence (symptoms recur post-antibiotics, regardless of culture results).
Duration of hospital stay (ICU/ general ward) | Through study completion, an average of 1 month
Proportion of patients with infections caused by antibiotic resistant bacteria | Through study completion, an average of 1 month
Direct medical costs of prescribed antibiotics, the assessment of serum procalcitonin (PCT assay) and hospital stay cost. | Through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Arjen Dondorp, Professor, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Chattogram Medical College Hospital (CMCH), Chittagong, Chattogram, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Participant data and results from blood analyses stored in the database may be shared according to the terms defined in the Mahidol Oxford Tropical Medicine Research Unit (MORU) data sharing policy with other researchers to use in the future. Datasets will be de-identified to ensure patient privacy and confidentiality.

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT05955612/SAP_001.pdf